CLINICAL TRIAL: NCT06684301
Title: Study on Predictive Factors, Safety and Efficacy of Endoscopic Retrograde Accessory Pancreatography in Chronic Pancreatitis: a Prospective Cohort Study
Brief Title: Study on Predictive Factors, Safety and Efficacy of Endoscopic Retrograde Accessory Pancreatography in CP
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHEC2022-238
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic Pancreatitis; Endoscopic Retrograde Pancreatography; Accessory Pancreatic Duct; Technical Success; Complication
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic pancreatitis (CP) can manifest characteristic pathological modifications such as pancreatic duct stenosis and pancreatic duct lithiasis. The endoscopic access to the main pancreatic duct through the major duodenal papilla is prevalently recognized as the most preponderant approach for endoscopic treatment of CP. Given that a multitude of CP patients are accompanied by main pancreatic duct stricture and distortion, certain patients encounter failure in main papilla angiography or are unable to achieve deep cannulation of the pancreatic duct, thus necessitating endoscopic retrograde accessory pancreatic ductography via the accessory papilla to augment the success rate of endoscopic drainage. Presently, there lacks a large - scale case report concerning the proportion of patients receiving main and accessory pancreatic ductography treatment and the safety and efficacy of endoscopic retrograde accessory pancreatic ductography in the treatment of CP. This study endeavors to establish a prospective cohort to document the proportion of CP patients undergoing main and accessory pancreatic duct angiography treatment and their clinical features during the initial endoscopic retrograde pancreatography (ERP). The main analysis centers on identifying the predictive factors for resorting to accessory pancreatic duct treatment subsequent to the failure of primary pancreatic duct angiography and assessing the safety and efficacy of endoscopic retrograde accessory pancreatic ductography in the treatment of CP.

DETAILED DESCRIPTION:
In recent years, with the development of endoscopic retrograde cholangiopancreatography (ERCP) technology, therapeutic ERCP has emerged as a first - line therapeutic modality for CP owing to its advantages of minimal invasiveness and high-level safety. The endoscopic access to the main pancreatic duct through the major duodenal papilla is commonly recognized as the preponderant approach for endoscopic treatment of CP. Nevertheless, in clinical practice, it has been observed that in a portion of CP patients, due to pancreatic divisum, distortion or stricture of the main pancreatic duct or other reasons, either the main papilla angiography fails or deep cannulation of the pancreatic duct cannot be achieved, thereby necessitating endoscopic retrograde accessory pancreatic ductography via the minor papilla. Previously, two small-sample retrospective studies analyzed the scenarios where CP patients with main pancreatic duct obstruction resulting from calculi, stenosis, etc. required attempts at accessory pancreatic ductography. The results demonstrated favorable safety and efficacy of accessory pancreatic duct treatment. In this prospective study, CP patients undergoing ERP for the first time in the pancreatic disease area of the Gastroenterology Department of Changhai Hospital were enrolled. After routine main papilla angiography, those with failed treatment via the main pancreatic duct were subjected to an attempt at endoscopic retrograde accessory pancreatic ductography through the minor papilla. Based on the distinct endoscopic retrograde angiography modalities and treatment outcomes in clinical practice, different subgroups were established. The number of cases receiving treatment via the main and accessory pancreatic ducts was tallied respectively. The clinical features of CP patients with successful main pancreatic duct drainage and those with failed drainage were compared. Emphasis was placed on analyzing the predictive factors for CP patients with failed main pancreatic duct angiography who then attempted accessory pancreatic duct angiography, as well as evaluating the safety and clinical efficacy of endoscopic retrograde accessory pancreatic ductography in CP patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pancreatitis hospitalized in Changhai Hospital from 2022.09.15 to 2024.01.18.
* Patients who completed endoscopic retrograde pancreatography.
* Aged 18 to 70 years,male or female.

Exclusion Criteria:

* Patients who accepted endoscopic retrograde pancreatography before.
* History of pancreatic surgery or Billroth II gastrectomy.
* Acute pancreatitis exacerbation or acute exacerbation of chronic pancreatitis
* Panceratic benign or malignant tumors.
* Pregnant or breastfeeding women.
* Patients who refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Changhai Hospital from 2022.09.15 to 2024.01.18.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
Success rate of accessory pancreatic ductography. | during ERCP procedure
  The success rate of accessory pancreatic ductography is the percentage of successful imaging operations of the accessory pancreatic duct, crucial for assessing the efficacy of relevant procedures.

SECONDARY OUTCOMES:
post-ERCP complications | 30 days after ERCP procedure
  Major post-ERCP complications includes post-ERCP pancreatitis, bleeding, infection, and perforation, which are classified as mild, moderate, or severe, depending mainly on the length of hospitalization and the need for invasive treatment.
clearance rates of pancreatic duct stones | during ERCP procedure
  Clearance rates have been defined as complete, partial, or failure if the proportion of stones cleared was > 90%, 50% - 90%, or < 50%, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tringali A, Voiosu T, Schepis T, Landi R, Perri V, Bove V, Voiosu AM, Costamagna G. Pancreas divisum and recurrent pancreatitis: long-term results of minor papilla sphincterotomy. Scand J Gastroenterol. 2019 Mar;54(3):359-364. doi: 10.1080/00365521.2019.1584640. Epub 2019 Mar 17. PMID 30880501
- [Background] Brown NG, Howell DA, Brauer BC, Walker J, Wani S, Shah RJ. Minor papilla endotherapy in patients with ventral duct obstruction: identification and management. Gastrointest Endosc. 2017 Feb;85(2):365-370. doi: 10.1016/j.gie.2016.07.066. Epub 2016 Aug 13. PMID 27530069
- [Background] Kwon CI, Gromski MA, Sherman S, El Hajj II, Easler JJ, Watkins J, McHenry L, Lehman GA, Fogel EL. Clinical response to dorsal duct drainage via the minor papilla in refractory obstructing chronic calcific pancreatitis. Endoscopy. 2017 Apr;49(4):371-377. doi: 10.1055/s-0042-120996. Epub 2017 Feb 15. PMID 28201840
- [Background] Moffatt DC, Cote GA, Avula H, Watkins JL, McHenry L, Sherman S, Lehman GA, Fogel EL. Risk factors for ERCP-related complications in patients with pancreas divisum: a retrospective study. Gastrointest Endosc. 2011 May;73(5):963-70. doi: 10.1016/j.gie.2010.12.035. Epub 2011 Mar 9. PMID 21392753